CLINICAL TRIAL: NCT06748547
Title: Effects of Scalp Nerve Block on Postoperative Pain, Hemodynamics and Surgical
Brief Title: Effects of Scalp Nerve Block on Postoperative Pain, Hemodynamics and Surgical Stress Response in Craniotomy Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Head of Anesthesia and reanimation, Umraniye Education and Research Hospital
Other Study IDs: UERH-AR-ZT-10
Record Dates: First submitted 2024-10-10; First posted 2024-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Analgesia; Post Operative Pain
Keywords: scalp nerve block,Craniotomy,postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Group pre-incisional: received 0.5% 20 ml bupivacaine preincisional before the nail head was placed
  Interventions: Procedure: scalp nerve block
- 2: Group post-incisional: received 0.5% 20 ml bupivacaine postcisional after the skin incision was closed
  Interventions: Procedure: scalp nerve block

INTERVENTIONS:
Procedure: scalp nerve block — scalp nerve block is performed bilaterally by an anesthesiologist after induction of anesthesia and 5 minutes before head immobilization, according to the technique described by Pinosky et al. Prepare a syringe (20 mL) for scalp blocks. It is performed using 0.35% bupivacaine and 5 mcg epinephrine (1:2,000,000) using a 23-gauge needle inserted at a 45° angle to the skin and penetrating deeply into the outer edge of the scalp.

SUMMARY:
The hypothesis of this study is that preincisional scalp nerve block will reduce postoperative opioid use and surgical stress response compared to postincisional scalp nerve block in craniotomy surgery with general anesthesia.

DETAILED DESCRIPTION:
Craniotomy is an effective treatment method for cerebral diseases and injuries, and postoperative pain is an important clinical problem. The most painful stages of craniotomy are the placement of a nail head and skin incision. Therefore, in these stages, it is necessary to increase the depth of anesthesia with additional analgesic administration to prevent hemodynamic responses such as tachycardia and hypertension. In patients with impaired cerebral autoregulation, a sudden increase in systemic blood pressure can cause a sudden increase in intracranial pressure, which accelerates intracranial hypertension. High oxygen consumption and catecholamine release caused by postoperative pain can lead to increased cerebral perfusion and increased intracranial pressure, which can predispose to intracranial hematoma. Effective postoperative pain management is important to prevent these systemic changes, improve rehabilitation, and improve long-term outcomes.

In addition, early postoperative pain management can prevent the development of central sensitization and chronic pain caused by surgical tissue damage.

In recent years, studies aimed at controlling postoperative pain starting from the preoperative period have brought the concept of preemptive analgesia to the agenda. Preemptive analgesia is applied before the painful stimulus in order to reduce the pain. Studies have suggested that surgical trauma causes an increase in nociceptive afferent transmission and causes changes in the excitation threshold in both peripheral and central neurons, and it is thought that postoperative pain can be controlled by preoperative blockade of this mechanism. Multimodal analgesia includes the use of single agents in postoperative pain control, especially the use of different pain control mechanisms to reduce the opioid dose, improve the analgesic effect and minimize the risk of side effects.

Scalp nerve block (SSB) is widely used to reduce hemodynamic response and incisional pain during craniotomy. Analgesia can be achieved by blocking the greater and lesser occipital nerves, supraorbital and supratrochlear nerves, zygomatico-temporal nerve, auriculo-temporal nerve and greater auricular nerve. SBB is combined with non-opioid drugs with different mechanisms of action to maximize the analgesic effect. Traumatic stimulation, such as surgery, acts on peripheral nerve pain receptors and produces nerve impulses that are transmitted to spinal dorsal horn neurons via Aδ and C fibers, and pain occurs after loading and integration. SSB can interrupt this pathway. Effective postoperative analgesia can reduce complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-65
* ASA 1-3 score

Exclusion Criteria:

* Chronic hypertension
* Arrhythmia
* body mass index (BMI) over 40 kg/m2
* Bleeding diathesis
* Allergy
* Serious cardiovascular, pulmonary, renal and hepatic disease
* Local infection at the injection site
* Alcohol and substance abuse
* Neurological sequelae, mental retardation
* GCS under 15
* Patients admitted to the intensive care unit as intubated
* Pregnancy
* Those with a history of chronic pain
* Scalp infection
* Use of vozoactive drugs
* Patients with previous craniotomy
* Patients who do not accept

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo cranitomy with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
hemodynamic parameters | 24 hours
  mean arterial pressure (mmHg)

SECONDARY OUTCOMES:
amount of opioid received during surgery | 24 hours
  remifentanil total dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No